CLINICAL TRIAL: NCT04534530
Title: Does Screening of Coronary Artery Disease an Efficient Public Health Strategy in Patients With Type 2 DIABetes at Very High Cardiovascular Risk: Target Trial Emulation From the National Healthcare System Claims Databases in France
Brief Title: Does Screening of Coronary Artery Disease an Efficient Public Health Strategy in Patients With Type 2 DIABetes
Acronym: SCADIAB
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/68
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cost / efficiency ratio; French health data base; Ischemic heart disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: The experimental group "systematic screening for ischemic heart disease" will be identified during the screening period by performing at least one systematic screening examination, regardless of the frequency, for ischemic heart disease in patients. diabetics at very high cardiovascular risk, without known coronary heart disease, by at least one non-invasive functional cardiovascular exploration outside the resting ECG.
  Interventions: Other: Systematic screening for ischemic heart disease in type 2 diabetic patients
- Control: The control group "Absence of systematic screening for ischemic heart disease" will be identified during the pre-selection period by the absence of a non-invasive functional cardiovascular exploration (examinations mentioned above) in T2D with very high cardiovascular risk, with no known coronary heart disease, apart from performing a resting ECG
  Interventions: Other: Systematic screening for ischemic heart disease in type 2 diabetic patients

INTERVENTIONS:
Other: Systematic screening for ischemic heart disease in type 2 diabetic patients — Systematic screening for ischemic heart disease in type 2 diabetic patients at very high cardiovascular risk, without known coronary heart disease.

SUMMARY:
The purpose of SCADIAB is to assess the real-life efficiency of systematic screening for ischemic heart disease in T2DM patients at very high cardiovascular risk, without known coronary heart disease, from the databases of the National Health Data System (SNDS).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is associated with an increased risk of cardiovascular and overall mortality. Cardiovascular disease is the leading cause of death, primarily ischemic heart disease, which is often early and can occur in asymptomatic diabetic patients, hence the potential benefit of routine screening to improve their cardiovascular prognosis.

There is a notable disparity between the recommendations of the french High Authority of Health (HAS) and those of learned societies. The HAS does not recommend routine screening for silent ischemic heart disease in all asymptomatic T2DM patients without known coronary heart disease, apart from a resting electrocardiogram (ECG). Functional cardiovascular examinations should be reserved for situations of high cardiovascular risk, particularly the presence of history, clinical symptoms or ECG abnormalities in favor of cardiovascular disease. On the other hand, the main learned societies of diabetology and cardiology recommend systematic screening for silent ischemic heart disease in a larger T2DM population (age> 60 years, duration of diabetes> 10 years and at least 2 cardiovascular risk factors). In terms of current clinical practice, a majority of physicians prescribe screening for silent ischemic heart disease in diabetic patients by functional examinations (stress test, myocardial tomoscintigraphy coupled with a stress test, stress echocardiography) . The investigators carried out two surveys with fellow cardiologists and diabetologists in Bordeaux and at the national level which confirm this frequent practice of screening.

The level of scientific evidence currently seems sufficient not to recommend systematic screening for silent ischemic heart disease in all diabetic patients. Four main randomized and controlled studies have not shown any benefit from this screening in terms of reducing major cardiovascular events in all T2DM patients. However, doubt remains in T2DM patients at very high cardiovascular risk, who may benefit from this strategy, but in whom no studies have been performed to date.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 40 years (on 2015/01/01),
* T2DM (ALD or hospitalization for T2DM or at least 3 deliveries of at least one oral or injectable anti-diabetic drug over a year (or 2 deliveries in the event of quarterly conditioning) without ALD or hospitalization for type 1 diabetes, secondary diabetes or diabetes gestational),
* Duration of diabetes greater than or equal to 7 years (the data available in the SNDS do not allow for an inclusion criterion of duration of diabetes> 7 years) (identified in 2008),
* Patients with regular follow-up by a doctor (GP, cardiologist, endocrinologist) defined as having at least one contact per year (during the pre-selection period),
* Affiliated with the general health insurance scheme,
* With at least 2 cardiovascular risk factors: obesity (hospitalization for obesity or at least 3 deliveries of an anti-obesity drug over one year), high blood pressure (hospitalization for high blood pressure or at least 3 deliveries of at least one antihypertensive medication over one year), hypercholesterolemia (at least 3 prescriptions for statin and / or ezetimibe), or chronic obstructive pulmonary disease (used as an indicator of chronic tobacco poisoning; ALD or hospitalization for chronic obstructive pulmonary disease),
* And presenting at least one of the following organ damage (during the pre-selection period): a) Carotid stenosis (hospitalization for carotid stenosis or act of carotid revascularization); b) AIT (ALD or hospitalization for AIT); c) Stroke (ALD or hospitalization for stroke); d) Arteriopathy obliterating of the lower limbs (ALD or hospitalization for arteriopathy obliterating of the lower limbs); e) Chronic renal disease (ALD or hospitalization for diabetic nephropathy, chronic renal failure or recourse to a technique of replacement or renal transplantation); f) Severe diabetic retinopathy treated by laser photocoagulation (ALD or hospitalization for diabetic retinopathy associated with an act of laser photocoagulation); g) Peripheral or autonomic diabetic neuropathy (ALD or hospitalization for diabetic peripheral or autonomic neuropathy),
* Alive on 2015/01/01.

Exclusion Criteria:

* Gestational diabetes,
* Secondary diabetes,
* Presence of ischemic heart disease (history or current disease): acute coronary syndrome, angina pectoris, unstable angina, or coronary revascularization,
* Visit to an emergency department for chest pain followed by admission to an intensive care unit for cardiology,
* Patients who have undergone one or more systematic screening examinations during the pre-selection phase.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the 3.3 million people treated pharmacologically for diabetes mellitus in France, at least 3 million would be T2DM. It can be assumed that at least 2.4 million are free from coronary heart disease. This survey also shows that arterial hypertension and dyslipidemia (the two main cardiovascular risk factors) are present respectively in 58% and 57% of T2DM patients, and renal, neuropathic, or retinal complications are present respectively in 10%, 11% and 8% of them. Therefore, it can be estimated that at least 90,000 T2DM patients would be eligible (at least 2 cardiovascular risk factors and one other vascular disease) to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness analysis of routine screening for ischemic heart disease in T2DM patients | 4 years after inclusion
  The cost-effectiveness analysis is based on the differential cost per year of life gained at 4 years from the point of view of Health Insurance (SNDS).

SECONDARY OUTCOMES:
Cost/consequence analysis for ischemic heart disease in T2DM patients. | 4 years after inclusion
  Direct costs (€) observed over 4 years for each strategy evaluated (screening and no screening ischemic heart disease). Based on SNDS analysis.
Budget impact analysis for Health Insurance of the most efficient strategy | 4 years after inclusion
  Net benefit for Health Insurance (€) from promoting the most efficient strategy: screening or no screening ischemic heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Julien BEZIN, Dr, Study Chair — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — USMR
Locations (1):
- Hopital Haut-Leveque, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammedi K, Preaubert N, Cariou T, Rigalleau V, Foussard N, Piazza L, Bairras-Martin C, Couffinhal T, Bezin J, Benard A. Cost-effectiveness of screening of coronary artery disease in patients with type 2 DIABetes at a very high cardiovascular risk (SCADIAB study) rational and design. Cardiovasc Diabetol. 2021 Mar 13;20(1):63. doi: 10.1186/s12933-021-01253-2. PMID 33714278